CLINICAL TRIAL: NCT00642876
Title: Investigation of the PRESTIGE® Cervical Disc Device at a Single Level for Symptomatic Cervical Disc Disease
Brief Title: PRESTIGE® Cervical Disc Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRESTIGE®
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Degenerative Cervical Disc Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): The Control cohort are patients that receive the fusion treatment.
  Interventions: Device: Allograft Fusion and ATLANTIS™ Cervical Plate System
- Investigational (Experimental): The Investigational cohort are the study patients that received the PRESTIGE® Cervical Disc.
  Interventions: Device: PRESTIGE® Cervical Disc

INTERVENTIONS:
Device: Allograft Fusion and ATLANTIS™ Cervical Plate System — The patients that received the control treatment underwent a single level anterior cervical fusion procedure involving allograft bone and the ATLANTIS™ Cervical Plate System.
  Other Names: ATLANTIS™
  Arms: Control
Device: PRESTIGE® Cervical Disc — The PRESTIGE® Cervical Disc is a stainless steel device that was inserted into the intervertebral disc space. The device is composed of two metal plates that interface via a ball and socket mechanism permitting segmental spinal motion.
  Other Names: PRESTIGE®
  Arms: Investigational

SUMMARY:
The purpose of this clinical investigation is to evaluate the safety and effectiveness of the ACD in the single level surgical treatment of patients with symptomatic cervical degenerative disc disease. The primary follow-up information obtained from this clinical investigation are used to support a PMA application for the ACD.

ELIGIBILITY:
Inclusion Criteria:

All patients participating in this study must meet all of the following inclusion criteria:

1. Cervical degenerative disc disease defined as:

   intractable radiculopathy and/or myelopathy with at least one of the following items producing symptomatic nerve root and/or spinal cord compression which is documented by patient history (e.g., neck and/or arm pain], functional deficit, and/or neurological deficit, and radiographic studies (e.g., CT, MRI, x-rays, etc).
   1. herniated disc;
   2. osteophyte formation;
2. One cervical level requiring surgical treatment;
3. C3-C4 disc to C6-C7 disc level of involvement;
4. Unresponsive to non-operative treatment for approximately six weeks or has the presence of progressive symptoms or signs of nerve root/spinal cord compression in the face of continued non-operative management;
5. No previous surgical intervention at the involved level or any subsequent, planned/staged surgical procedure at the involved or adjacent level(s);
6. Is at least 18 years of age, inclusive, at the time of surgery;
7. Preoperative Neck Disability Index score > or = 30;
8. Has a preoperative neck pain score of > 20 based on the Preoperative Neck and Arm Pain Questionnaire.
9. If of child-bearing potential, patient is not pregnant at the time of surgery;
10. Is willing to comply with the study plan and sign the Patient Informed Consent Form.

Exclusion Criteria:

A patient meeting any of the following criteria is to be excluded from the study:

1. Has a cervical spinal condition other than symptomatic cervical disc disease requiring surgical treatment at the involved level;
2. Documented or diagnosed cervical instability defined by dynamic (flexion/extension) radiographs showing:

   1. Sagittal plane translation > 3.5 mm or;
   2. Sagittal plane angulation > 20.
3. More than one cervical level requiring surgical treatment;
4. Has a fused level adjacent to the level to be treated;
5. Has severe pathology of the facet joints of the involved vertebral bodies;
6. Previous surgical intervention at the involved level;
7. Has been previously diagnosed with osteopenia or osteomalacia;
8. Has any of the following that may be associated with a diagnosis of osteoporosis (if Yes to any of the below risk factors, a DEXA Scan will be required to determine eligibility):

   1. Postmenopausal Non-Black female over 60 years of age and weighs less than 140 pounds.
   2. Postmenopausal female that has sustained a non-traumatic hip, spine, or wrist fracture.
   3. Male over the age of 70.
   4. Male over the age of 60 that has sustained a non-traumatic hip or spine fracture.

   If the level of BMD is a T score of -3.5 or a T score of -2.5 with vertebral crush fracture, then the patient is excluded from the study.
9. Has presence of spinal metastases;
10. Has overt or active bacterial infection, either local or systemic;
11. Has severe insulin dependent diabetes;
12. Has chronic or acute renal failure or prior history of renal disease;
13. Has fever (temperature > 101 F oral) at the time of surgery;
14. Has a documented allergy or intolerance to stainless steel, titanium, or a titanium alloy;
15. Is mentally incompetent. (If questionable, obtain psychiatric consult);
16. Is a prisoner;
17. Is pregnant;
18. Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug abuse;
19. Has received drugs which may interfere with bone metabolism within two weeks prior to the planned date of spinal surgery (e.g., steroids or methotrexate), excluding routine perioperative anti-inflammatory drugs;
20. Has a history of an endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's Disease, renal osteodystrophy, Ehlers-Danlos Syndrome, or osteogenesis imperfecta);
21. Has a condition that requires postoperative medications that interfere with the stability of the implant or fusion, such as steroids. (This does not include low dose aspirin for prophylactic anticoagulation and routine perioperative anti-inflammatory drugs);
22. Has received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the16 weeks following Artificial Cervical Disc implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2002-10; Primary Completion 2006-07 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is overall success, which consists of NDI score, neuro status success, with/without FSU disc ht success, no serious AE classified as "implant/surgical procedure associated", and no secondary surgical procedure classified as failure | 24 months

SECONDARY OUTCOMES:
The secondary outcomes are radiographic success, medical outcomes SF-36 patient survey (MCS & PCS) success, neck pain status, arm pain status, patient satisfaction, patient global perceived effect, gait assessment, foraminal compression test | 24 months

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - North Alabama Neurological, Huntsville, Alabama
  - Montgomery Neurosurgical, Montgomery, Alabama
  - University of California, Davis, Sacramento, California
  - The Spine Institute, Santa Monica, California
  - Orlando Neurosurgery, Winter Park, Florida
  - Atlanta Brain and Spine Care, Atlanta, Georgia
  - Emory Orthop and Spine Center, Atlanta, Georgia
  - Hughston Clinic, Columbus, Georgia
  - Central Illinois Neuroscience, Bloomington, Illinois
  - Loyola University Medical Center, Oak Park, Illinois
  - Orthoindy, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Baton Rouge Orth Clinic, Baton Rouge, Louisiana
  - Neurosurgery Ass, P.A., Baltimore, Maryland
  - Michigan Brain & Spine Institute, Ypsilanti, Michigan
  - The Ortho Center of St. Louis, Chesterfield, Missouri
  - Springfield Neurological Institute, Springfield, Missouri
  - Surgical Neurology New Hampshire Neurospine Institute, Bedford, New Hampshire
  - Buffalo Neurosurgery Group, West Seneca, New York
  - Oregon Health & Science University, Portland, Oregon
  - Westphal Group, Lancaster, Pennsylvania
  - Center of Neurosciences Orthopedics & Spine, P.C., Dakota Dunes, South Dakota
  - Spine Surgery Associates, Chattanooga, Tennessee
  - Semmes Murphey, Memphis, Tennessee
  - Howell Allen Clinic, Nashville, Tennessee
  - Brain and Spine Center of Texas, Plano, Texas
  - Neurosugical Associates, PC, Richmond, Virginia
  - Inland Neurosurgery & Spine Associates, P.S., Spokane, Washington
  - University of Wisconsin Medical School, Madison, Wisconsin
  - Central Wyoming Neurosurgery, Casper, Wyoming
  - Wyoming Brain and Spine Institute, Casper, Wyoming

REFERENCES:
- [Background] Burkus JK, Haid RW, Traynelis VC, Mummaneni PV. Long-term clinical and radiographic outcomes of cervical disc replacement with the Prestige disc: results from a prospective randomized controlled clinical trial. J Neurosurg Spine. 2010 Sep;13(3):308-18. doi: 10.3171/2010.3.SPINE09513. PMID 20809722
- [Background] Mummaneni PV, Burkus JK, Haid RW, Traynelis VC, Zdeblick TA. Clinical and radiographic analysis of cervical disc arthroplasty compared with allograft fusion: a randomized controlled clinical trial. J Neurosurg Spine. 2007 Mar;6(3):198-209. doi: 10.3171/spi.2007.6.3.198. PMID 17355018
- [Derived] Gornet MF, Lanman TH, Burkus JK, Hodges SD, McConnell JR, Dryer RF, Schranck FW, Copay AG. One-Level Versus 2-Level Treatment With Cervical Disc Arthroplasty or Fusion: Outcomes Up to 7 Years. Int J Spine Surg. 2019 Dec 31;13(6):551-560. doi: 10.14444/6076. eCollection 2019 Dec. PMID 31970051
- [Derived] Arnold PM, Anderson KK, Selim A, Dryer RF, Kenneth Burkus J. Heterotopic ossification following single-level anterior cervical discectomy and fusion: results from the prospective, multicenter, historically controlled trial comparing allograft to an optimized dose of rhBMP-2. J Neurosurg Spine. 2016 Sep;25(3):292-302. doi: 10.3171/2016.1.SPINE15798. Epub 2016 Apr 29. PMID 27129045
- [Derived] Burkus JK, Traynelis VC, Haid RW Jr, Mummaneni PV. Clinical and radiographic analysis of an artificial cervical disc: 7-year follow-up from the Prestige prospective randomized controlled clinical trial: Clinical article. J Neurosurg Spine. 2014 Oct;21(4):516-28. doi: 10.3171/2014.6.SPINE13996. Epub 2014 Jul 18. PMID 25036218